CLINICAL TRIAL: NCT04178863
Title: Efficacy of Topical Latanoprost 0.005% Verses Timolol 0.5% Demonstrated by Corneal Biomechanical Correcting Modified Goldmann Prism
Brief Title: CATS Tonometer IOP Reduction Latanoprost Verses Timolol
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Intuor Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019004
Record Dates: First submitted 2019-11-23; First posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Glaucoma; Drugs
MeSH Terms: conditions — Glaucoma | interventions — Latanoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- lataprost (Active Comparator): latanoprost use
  Interventions: Device: CATS Tonometer
- timolol (Active Comparator): timolol group
  Interventions: Device: CATS Tonometer; Drug: Latanoprost

INTERVENTIONS:
Device: CATS Tonometer — latanoprost vs. timolol
  Other Names: latanoprost v. timolol
Drug: Latanoprost — latanoprost IOP reduction
  Arms: timolol

SUMMARY:
Topical Prostaglandin Analog vs Betablocker - Corneal Biomechanical Evaluation using CATS Tonometer Prism

DETAILED DESCRIPTION:
This clinical trial is a prospective, controlled, study and will be performed at one clinical investigative site in Tucson Arizona1. The purpose of this study is to determine if the device, CATS tonometer prism, measures intraocular pressure significantly differently than the current standard of care tonometer prism (Goldmann) before and after institution of topical prostaglandin analogs (PGA) for glaucoma treatment. Fifty percent of patients will be randomly placed on topical beta blockers as a control. The difference PGAs and beta blockers would be a measurement of the amount of corneal biomechanical changes made due to the PGA controlled for the effect of IOP lowering by the beta -blocker group.

ELIGIBILITY:
Inclusion Criteria:

* • Male and female patients, at least 18 years of age

  * Subject has a clear understanding and agrees to all the conditions of the informed consent form

Exclusion Criteria:

* Subjects shall be selected in accordance with the following exclusion criteria

  * Subject has undergone ocular surgery within the last 3 months
  * Uncontrolled systemic disease that in the opinion of the Investigator would put the subject's heath at risk
  * Pregnant or nursing women
  * Those who have had corneal surgery including corneal laser surgery
  * Microphthalmos
  * Buphthalmos
  * Severe Dry eyes
  * Lid squeezers - blepharospasm
  * Nystagmus
  * corneal or conjunctival infection.

Ages: 18 Years to 101 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
IOP reduction | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona Eye Consultants, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Radcliffe N, Berdahl J, Ibach M, Schweitzer J, Levine J, McCafferty S. Improved Efficacy of Topical Latanoprost 0.005% Demonstrated by Corneal Biomechanical Correcting Modified Goldmann Prism. Clin Ophthalmol. 2020 Aug 10;14:2245-2253. doi: 10.2147/OPTH.S264055. eCollection 2020. PMID 32884231